CLINICAL TRIAL: NCT05641272
Title: Prospective, Randomised, DBPC Clinical Trial to Evaluate the Efficacy and Safety of Polymerized and Mannan Conjugated Allergen Extract of Dermatophagoides for the Treatment of Allergic Rhinitis/Rhinoconjunctivitis With or Without Asthma
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Polymerized, Mannan-Conjugated Dermatophagoides Allergen Extract
Acronym: MM09-SLIM
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Collaborators: LAT Research (Other); Xolomon Tree S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MM09-SLG-056
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-11

CONDITIONS: Allergic Rhinitis; Allergic Asthma; Allergic Rhinoconjunctivitis; Allergy to House Dust Mite
Keywords: Allergy; Mites; Hypersensitivity; Rhinitis; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Dust Mite Allergy; Hypersensitivity; Rhinitis

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the trial, both the investigator and the subjects included will be unaware of the treatment each subject is receiving.
  Blinding is intended to minimize potential biases resulting from differences in treatment or assessment of subjects. It is also intended to reduce as much as possible the interpretation of the results that could arise as a consequence of the investigator or the subject knowing the assigned treatment.
  The person in charge of data analysis will also not know the treatment assigned to each subject until the database has been closed.
  So that neither the subject nor the investigator will know which treatment each subject is receiving, all trial medication will be identical in outer packaging and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: sublingual allergoid-mannan conjugates (MM09 at 3.000 UTm/mL) (Experimental): Allergoid (Dermatophagoides pteronyssinus and Dermatophagoides farinae)-mannan conjugates (MM09) at 3.000 UTm/mL for sublingual immunotherapy. The dose is 2 sprays daily applied to the sublingual mucosa for 6 months.
  Interventions: Biological: 3,000 MM09
- Group II: sublingual allergoid-mannan conjugates (MM09 at 9.000 UTm/mL) (Experimental): Allergoid (Dermatophagoides pteronyssinus and Dermatophagoides farinae)-mannan conjugates (MM09) at 9.000 UTm/mL for sublingual immunotherapy.. The dose is 2 sprays daily applied to the sublingual mucosa for 6 months.
  Interventions: Biological: 9,000 MM09
- Group III: sublingual placebo (Placebo Comparator): The same solution, presentation, method of administration, frequency, and duration as the active treatment, but without active ingredients.The dose is 2 sprays daily applied to the sublingual mucosa for 6 months.
  Interventions: Other: Placebo sublingual

INTERVENTIONS:
Biological: 3,000 MM09 — Allergoid (Dermatophagoides pteronyssinus and Dermatophagoides farinae)-mannan conjugates (MM09) at 3.000 UTm/mL for sublingual immunotherapy.
  Arms: Group I: sublingual allergoid-mannan conjugates (MM09 at 3.000 UTm/mL)
Biological: 9,000 MM09 — Allergoid (Dermatophagoides pteronyssinus and Dermatophagoides farinae)-mannan conjugates (MM09) at 9.000 UTm/mL for sublingual immunotherapy.
  Arms: Group II: sublingual allergoid-mannan conjugates (MM09 at 9.000 UTm/mL)
Other: Placebo sublingual — The same solution, presentation, method of administration, frequency, and duration as the active treatment, but without active ingredients.
  Arms: Group III: sublingual placebo

SUMMARY:
Prospective, randomised, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of polymerized and mannan conjugated allergen extract of Dermatophagoides for the treatment of allergic rhinitis/rhinoconjunctivitis with or without asthma.

The main objective of the clinical trial is to evaluate the clinical efficacy of the investigational medicinal product, administered sublingually, compared to placebo for the treatment of moderate-severe rhinitis/rhinoconjunctivitis with or without mild to moderate asthma and controlled using the Rhinitis/Rhinoconjunctivitis Combined Symptom and Medication Score (R-CSMS).

DETAILED DESCRIPTION:
Allergen-specific immunotherapy (AIT) has been shown to be effective in relieving symptoms, reducing medication use, and improving quality of life in patients with respiratory allergies). This is thought to be due to the induction of a state of tolerance to specific allergens with long-lasting effects after discontinuation of treatment. And it is accepted that immunotherapy is the only available method for allergists to improve or cure, partially or definitely, an allergic process The study population of this clinical trial will comprise subjects allergic to mites (Dermatophagoides pteronyssinus and/or D. farinae) with symptoms of moderate-severe rhinitis/rhinoconjunctivitis with or without mild to severe controlled asthma, suitable to allergen immunotherapy.

The primary efficacy endpoint will be the combined rhinitis/rhinoconjunctivitis symptom and medication score.

Every single day from the beginning of the administration of the investigational drug (V2-VF), the subject will be asked to score and register his/her symptoms and record medication consumption in an electronic diary following the instructions of the application. This diary will provide the symptom score and medication consumption for each subject during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form.
2. Male or female, aged between 12 and 60 years, both included.
3. Confirmed clinical history of inhalation allergy with moderate-severe rhinitis/rhinoconjunctivitis according to the ARIA classification with or without controlled mild-moderate intermittent or persistent asthma according to the definition of GEMA 5.0 y GINA caused by allergy to mites (D. pteronyssinus and/or D. farinae). The asthma diagnostic will be valid up to 24 months prior to signing the informed consent form.
4. Combined Symptom and Medication Score for moderate to severe rhinitis/rhinoconjunctivitis (RCSMS) ≥ 1,8 out of 3.
5. Positive skin prick test (wheal major diameter ≥ 5 mm) to a standardized allergen extract of Dermatophagoides pteronyssinus and/or Dermatophagoides farinae. The results will be valid up to 12 months prior to signing the informed consent form.
6. Specific IgE against a complete extract of Dermatophagoides pteronyssinus and/or D. farinae or any the molecular components of allergenic sources with a value ≥ 3.5 kU/L. The results will be valid up to 12 months prior to signing the informed consent form.
7. Subjects shall preferably be monosensitised to the study allergens. In case of subjects sensitised to other aeroallergens, only those with the following characteristics may be included in the study (results will be valid up to 12 months prior to signing the informed consent form):

   * Subjects with a positive skin prick test to Blomia tropicalis and Lepidoglyphus destructor, whose wheal major diameter and specific IgE values do not exceed or equal the values for the study allergens.
   * Subjects with a positive skin prick test for dander if they have occasional exposure and symptoms.
   * Subjects with positive skin prick test to pollens, whose specific IgE values do not exceed or equal the values for the study allergens and who also do not have exacerbations during pollen season. The maximum specific IgE value to theses allergens is 17.5 kU/L.
8. Subjects with negative skin prick test to mold. In case specific IgE determination have been performed, the result must be <0.35 kU/L.
9. Women of childbearing age (since menarche) must present a negative urine pregnancy test at the time of trial enrollment.
10. Women of childbearing age must commit to using and adequate contraception method.
11. Subjects capable of complying with a dosage regimen.
12. Subjects owning a smartphone to register symptoms and medication consumption.

Exclusion Criteria:

1. Subjects polysensitized to other aeroallergens with clinically relevant symptoms.
2. Subjects who have received previous immunotherapy in the preceding 5 years to any of the tested allergens or a cross-reactive allergen or are currently receiving immunotherapy with any allergen.
3. Patients in whom immunotherapy may be subject to an absolute general contraindication according to the criteria of the Immunotherapy Committee of the Spanish Society of Allergy and Clinical Immunology and the European Allergy and Clinical Immunology Immunotherapy Subcommittee may not be included.
4. Subjects with uncontrolled severe asthma, and/or with FEV1 <80% of baseline despite adequate pharmacological treatment by the time of the enrolment.
5. Subjects on treatment with ß-blockers.
6. Subjects on treatment with immunosuppressive or biological drugs.
7. Subjects who are unstable by the time of enrolment (respiratory infection, febrile process, acute pruritus, etc.).
8. Subjects with chronic urticaria during the last 2 years, severe anaphylaxis or with hereditary angioedema history.
9. Subjects with any pathology in which the administration of adrenaline is contraindicating (hyperthyroidism, hypertension, heart disease, etc.) according to the investigator discretion.
10. Subjects with any other disease not related to moderate rhinoconjunctivitis or asthma, but potentially serious and that could interfere with treatment and follow-up (epilepsy, psychomotor disorders, diabetes, malformations, multi-surgery, nephropathy, etc.), according to the investigator discretion.
11. Subjects with severe autoimmune disease (thyroiditis, lupus, etc.), tumour diseases or diagnosed with immunodeficiencies.
12. Subject whose condition prevents him/her from offering cooperation and/or who presents severe psychiatric disorders, according to the investigator discretion.
13. Subjects with known allergy to the other components of the investigational product other than allergen study.
14. Subjects with lower airway diseases other than asthma such as emphysema or bronchiectasis.
15. Pregnant or breastfeeding women.
16. Subjects who are immediate family members of researchers.
17. Concurrent participation in other clinical trials or previous participation within 30 days prior to inclusion.
18. History of severe systemic reactions, including food, hymenoptera venom, etc.
19. Subjects who have suffered a respiratory tract infection and/or asthma exacerbation within 4 weeks prior to screening.
20. Subjects with a history of significant renal disease or chronic liver disease.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rhinitis/rhinoconjunctivitis Combined Symptom and Medication Score (RCSMS) | 6 months
  Assessment of the number of rhinitis/rhinoconjunctivitis symptoms and medication consumption required to control these symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  Rhinitis/Rhinoconjunctivitis Combined Symptom and Medication Score will be based on the work done by Pfaar et al. The score for each rhinitis/rhinoconjunctivitis symptom will be 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe. Total daily symptom score = 0-3
  The score for Rhinitis/rhinoconjunctivitis medication will be: 0 = No medication; 1 = Oral or topical (eye or nose) non-sedating H1 antihistamines (H1A); 2 = Intranasal corticosteroids (INS) with/without H1A; 3 = Oral corticosteroids with/without (INS), with/without H1A. Total daily medication score = 0-3

SECONDARY OUTCOMES:
Rhinitis/ Rhinoconjunctivitis Symptom Score (RSS) | 6 months
  Assessment of the number of rhinitis/rhinoconjunctivitis symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for each rhinitis/rhinoconjunctivitis symptom will be 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe. Total daily symptom score = 0-3
Rhinitis/Rhinoconjunctivitis Medication Score (RMS) | 6 months
  Evaluation of the medication consumption required to control the rhinitis/rhinoconjunctivitis symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for rhinitis/rhinoconjunctivitis medication will be: 0 = No medication; 1 = Oral or topical (eye or nose) non-sedating H1 antihistamines (H1A); 2 = Intranasal corticosteroids (INS) with/without H1A; 3 = Oral corticosteroids with/without (INS), with/without H1A. Total daily medication score = 0-3
Asthma Combined Symptom and Medication Score (ACSMS) | 6 months
  Evaluation of the number of asthma symptoms and medication consumption required to control these symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for each asthma symptom will be: 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe. Total daily symptom score = 0-3
  The asthma medication will be scored based on the therapeutic step in which the drugs are included in the Guía Española para el Manejo del Asma (GEMA) 5.0 and Global Initiative for Asthma (GINA) 2020 guidelines. The scoring method is detailed in the article entitled "Combination of Allergic Asthma Symptom and Medication Scores in Allergen Immunotherapy Trials: A Proposal". Total daily medication score (ACSMS) = 0-3
Asthma Symptom Score (ASS) | 6 months
  Assessment of the number of asthma symptoms of each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for each asthma symptom will be: 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe. Total daily symptom score (ASS) = 0-3
Asthma Medication Score (AMS) | 6 months
  Evaluation of the medication consumption required to control the asthma symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  The medication will be scored based on the therapeutic step in which the drugs are included in the GEMA 5.0 and GINA 2020 guidelines. Total daily medication score (AMS) = 0-3
Asthma and Rhinitis/Rhinoconjunctivitis Symptom Score (ARSS) | 6 months
  Evaluation of the number of asthma and rhinitis/rhinoconjunctivitis symptoms of each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for each and asthma rhinitis/rhinoconjunctivitis symptom will be 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe. Total daily symptom score = 0-3
Asthma and Rhinitis/Rhinoconjunctivitis Medication Score (ARMS) | 6 months
  Assessment of the number of medication consumption required to control asthma and rhinitis/rhinoconjunctivitis symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for rhinitis/rhinoconjunctivitis medication will be: 0 = No medication; 1 = Oral or topical (eye or nose) non-sedating H1 antihistamines (H1A); 2 = Intranasal corticosteroids (INS) with/without H1A; 3 = Oral corticosteroids with/without (INS), with/without H1A.
  The asthma medication will be scored based on the therapeutic step in which the drugs are included in the GEMA 5.0 and GINA 2020 guidelines.
  Total daily medication score (ARMS) = 0-3
Asthma and Rhinitis/Rhinoconjunctivitis Combined Symptom and Medication Score (ARCSMS) | 6 months
  Evaluation of the number of asthma and rhinitis/rhinoconjunctivitis symptoms and medication consumption required to control these symptoms for each subject during the trial, for each group compared to the others, and compared to placebo.
  The score for each asthma and rhinitis / rhinoconjunctivitis symptom will be as follows: 0 = No symptoms; 1 = Mild; 2 = Moderate; 3 = Severe. Total daily symptom score = 0-3
  The score for rhinitis/rhinoconjunctivitis medication consumption will be: 0 = No medication; 1 = Oral or topical (eye or nose) non-sedating H1 antihistamines (H1A); 2 = Intranasal corticosteroids (INS) with/without H1A; 3 = Oral corticosteroids with/without (INS), with/without H1A. The score for the asthma medication will be based on the therapeutic step in which drugs are included in the GEMA 5 guide. Total daily medication score = 0-3
Symptom free-days (rhinitis/rhinoconjunctivitis, asthma) | 6 months
  Number of days that the subjects have no symptom
Medication free days (rhinitis/rhinoconjunctivitis, asthma) | 6 months
  Number of days that the subjects need no medication
Asthma exacerbations | 4 months
  Time elapsed to first asthma exacerbation, number, duration and severity.
Clinical benefit | 6 months
  Elapsed time to clinical benefit
Respiratory function | 6 months
  Forced expiratory volume at one second (FEV1) and peak expiratory flow (PEF) will be measured to assess the degree of airflow obstruction.
  International consensus guidelines suggest that in asthma the measurements of FEV1 and PEF are equivalent when expressed as the per cent of predicted values.
  FEV1 of 80 to 100 percent is generally considered normal. FEV1 between 60 and 79 percent of predicted indicates a mild obstruction FEV1 between 40 and 59 percent indicates a moderate obstruction
Number of eosinophil | 6 months
  A blood sampling will be performed determine the number of eosinophils.
Immunological parameters in blood | 6 months
  A blood sampling will be performed determine
  * Total immunoglobulin E (IgE)
  * Specific IgE and immunoglobulin G4 (IgG4)
  * Specific IgE/total IgE index
  * Immunoglobulin A (IgA )
  * Immunoglobulin G (IgG) anti-Saccharomyces cerevisiae (ASCA)(4)
Immunological parameters in nasal mucosa. | Month 2 and month 7
  A nasal sample will be taken using nasal swabs to determine the following immunological parameters:
  * Total and specific IgA
  * Total and specific IgG
Asthma Quality of Life Questionnaire (AQLQ) | Month 2 and month 7
  Asthma Quality of Life Questionnaire (AQLQ) consists of 32 items and 4 domains (symptoms, activity limitations, emotional function and environmental stimuli). Each item is scored from 1 ("no impairment") to 7 ("severe impairment")
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | 6 months
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) consists of 28 items (questions) and 7 domains (Activities, Sleep, General symptoms, Practical problems, Nose symptoms, Eye symptoms and Emotional).
  The score of each item for all domains, except for the emotional domain, ranges from 0 ("It did not bother me at all") to 6 ("It bothered me a lot"). The score for the emotional domain ranges from 0 ("Never") to 6 ("Always").
Asthma Control Questionnaire (ACQ 6) | 4 months
  The Asthma Control Questionnaire (ACQ-6) consists of 6 questions. In questions 1-6, subjects recall their experience over the past 7 days and respond using a 7-point scale from 0 ("totally controlled") to 6 ("extremely poorly controlled"). The score of the questionnaire is the mean of the 6 answers (i.e., the sum of the 6 answers divided by 6). The interpretation of the scores is as follows:
  * Less than or equal to 0.75: Adequate asthma control
  * From 0.75 to 1.50: Partially controlled asthma
  * Over 1.50: Inadequate asthma control
Asthma Control Questionnaire (ACQ 7) | 6 months
  The ACQ questionnaire consists of 7 questions (ACQ-7) In questions 1-6, patients recall their experience during the last 7 days and answer using a scale of 7 points (from 0 = fully controlled to 6 = extremely poorly controlled). The seventh question, which refers to the% FEV1 of the reference value, must be completed by an employee of the site. The questionnaire score is the mean of the 7 responses (ACQ-7)
  The interpretation of the scores is as follows:
  * Less than or equal to 0.75: Adequate control of asthma
  * From 0.75 to 1.50: Partially controlled asthma
  * More than 1.50: Inadequate asthma control
Visual Analogue Scales (VAS) | 7 months
  The visual analogue scale is a 10 cm straight line, where the left end means that the subject feels very bad, and the right end means that the subject feels very well. Throughout the trial, two VAS scale measurements will be used:
  * Subject's VAS, where the participant marks a dot on the line that matches his or her health status with respect to allergy symptoms.
  * Investigator's VAS, where the investigator must mark a dot on the line that matches the subject's health status with respect to allergy symptoms.
Consumption of health resources | 7 months
  For each subject, the number of times that due to allergy symptoms has done the following will be counted:
  * have visited the family doctor
  * have made an unscheduled visit to the specialist
  * has gone to the emergency room
  * has been hospitalized
  * have needed to contact the doctor by phone
Security parameters | Month 2 and month 7
  Global rate and severity of Adverse Events (AE) per administration and per subject
Number of Local Adverse Reactions | 6 months
  Local adverse reactions are those that appear at the site of the administration. They are classified into: Immediate (it appears during the first 30 minutes from the administration of investigational product) and Late (it appears after the first 30 minutes from the administration of investigational product)
Number of Systemic Adverse Reactions | 6 months
  Systemic adverse reactions are those that appear in other parts of the body other than the site of administration. Their severity will be classified according to World Allergy Organization, measured according to the following grades:
  * 1: Symptoms or signs present in a system/organ (cutaneous, Upper respiratory tract, Conjunctival or Other)
  * 2: Symptoms or signs of 2 or more organs systems listed in Grade 1
  * 3: Lower airway disease: Mild bronchospasm and/or Gastrointestinal/Abdominal cramps and/or vomiting/diarrhoea/Other Uterine cramps/Any symptoms/signs from grade 1 would be included.
  * 4: Lower airway: Severe bronchospasm not responding or worsening despite treatment and/or Upper airway/Laryngeal oedema with stridor /Any symptoms/signs from grades 1or 3 would be included.
  * 5: Lower or upper airway: Respiratory failure and/or Cardiovascular /Collapse/hypotension and/or Loss of consciousness (vasovagal excluded)/Any symptoms/signs from grades 1,3, or 4 would be included.
Number of Adverse Reactions to any medication | 7 months
  Number of Adverse Reactions to any medication administered for the treatment of AE/AR
Treatment adherence | 6 months
  At each visit, a new bottle shall be provided to the subject and the previous bottle shall be collected. The amount remaining in each returned bottle shall be analysed to assess adherence to treatment.
Compliance of the electronic diary | 6 months
  All subjects included in the trial will download the "ITK Diary Card" app on their mobile phone, which will be used as the subject's electronic diary. Subjects will fill in their symptoms and medication intake.
  At each visit, the investigator should review the subject's electronic diary to ensure compliance.
  For the calculation of the main variable, only those subjects that have reported data corresponding to at least 40% of the days will be considered. Therefore, for subjects with less than 40% of the reported data, the main variable cannot be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Fernando Maspero, MD, PhD, Principal Investigator — Fundación CIDEA
Locations (1):
- Fundación CIDEA, Buenos Aires, Paraguay, Argentina

REFERENCES:
- [Background] Malling HJ. The position of immunotherapy in the European Academy of Allergology and Clinical Immunology. J Investig Allergol Clin Immunol. 1997 Sep-Oct;7(5):356-7. No abstract available. PMID 9416545
- [Background] Sirvent S, Soria I, Cirauqui C, Cases B, Manzano AI, Diez-Rivero CM, Reche PA, Lopez-Relano J, Martinez-Naves E, Canada FJ, Jimenez-Barbero J, Subiza J, Casanovas M, Fernandez-Caldas E, Subiza JL, Palomares O. Novel vaccines targeting dendritic cells by coupling allergoids to nonoxidized mannan enhance allergen uptake and induce functional regulatory T cells through programmed death ligand 1. J Allergy Clin Immunol. 2016 Aug;138(2):558-567.e11. doi: 10.1016/j.jaci.2016.02.029. Epub 2016 Apr 13. PMID 27177779
- [Background] Soria I, Alvarez J, Manzano AI, Lopez-Relano J, Cases B, Mas-Fontao A, Canada FJ, Fernandez-Caldas E, Casanovas M, Jimenez-Barbero J, Palomares O, Vinals-Florez LM, Subiza JL. Mite allergoids coupled to nonoxidized mannan from Saccharomyces cerevisae efficiently target canine dendritic cells for novel allergy immunotherapy in veterinary medicine. Vet Immunol Immunopathol. 2017 Aug;190:65-72. doi: 10.1016/j.vetimm.2017.07.004. Epub 2017 Jul 23. PMID 28778325
- [Background] Nieto A, Mazon A, Nieto M, Ibanez E, Jang DT, Calaforra S, Alba P, Perez-Frances C, Llusar R, Montoro J, de Mateo A, Alamar R, El-Qutob D, Fernandez J, Moral L, Toral T, Anton M, Andreu C, Ferrer A, Flores IM, Cerda N, Del Pozo S, Caballero R, Subiza JL, Casanovas M. First-in-human phase 2 trial with mite allergoids coupled to mannan in subcutaneous and sublingual immunotherapy. Allergy. 2022 Oct;77(10):3096-3107. doi: 10.1111/all.15374. Epub 2022 May 27. PMID 35570712
- [Background] Pfaar O, Klimek L, Gerth van Wijk R. Clinically relevant outcome measures for new pharmacotherapy, allergen avoidance and immunotherapy trials in allergic rhinoconjunctivitis. Curr Opin Allergy Clin Immunol. 2015 Jun;15(3):197-203. doi: 10.1097/ACI.0000000000000164. PMID 25899694
- [Background] Caballero R, Grau A, Javaloyes G, Del Pozo S, Leon MA, Romero M, Casanovas M. Combination of Allergic Asthma Symptom and Medication Scores in Allergen Immunotherapy Trials: A Proposal. Int Arch Allergy Immunol. 2021;182(7):571-573. doi: 10.1159/000513543. Epub 2021 Jan 26. No abstract available. PMID 33498057
- [Background] Passalacqua G, Baena-Cagnani CE, Bousquet J, Canonica GW, Casale TB, Cox L, Durham SR, Larenas-Linnemann D, Ledford D, Pawankar R, Potter P, Rosario N, Wallace D, Lockey RF. Grading local side effects of sublingual immunotherapy for respiratory allergy: speaking the same language. J Allergy Clin Immunol. 2013 Jul;132(1):93-8. doi: 10.1016/j.jaci.2013.03.039. Epub 2013 May 15. PMID 23683513